CLINICAL TRIAL: NCT02728050
Title: Addition of Sorafenib to G-CSF, Cladribine, Cytarabine and Mitoxantrone (G-CLAM) in Adults With Newly-Diagnosed Acute Myeloid Leukemia (AML) Independent of FLT3-ITD Status: A Phase 1/2 Study
Brief Title: Filgrastim, Cladribine, Cytarabine, and Mitoxantrone With Sorafenib in Treating Patients With Newly-Diagnosed, Acute Myeloid Leukemia or High-Risk Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Bayer (Industry)
Responsible Party: Principal Investigator, Anna Halpern, Assistant Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9510; NCI-2016-00286 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9510 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1016000 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2016-03-14; First posted 2016-04-05 (Estimated); Results first posted 2023-06-29 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Acute Biphenotypic Leukemia; Acute Myeloid Leukemia; de Novo Myelodysplastic Syndrome; Myelodysplastic Syndrome; Myeloproliferative Neoplasm
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Myeloproliferative Disorders | interventions — Cladribine; Cytarabine; Filgrastim; Granulocyte Colony-Stimulating Factor; Mitoxantrone; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (sorafenib, G-CLAM) (Experimental): See Detailed Description.
  Interventions: Drug: Cladribine; Drug: Cytarabine; Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Drug: Mitoxantrone; Drug: Sorafenib

INTERVENTIONS:
Drug: Cladribine — Given IV
  Other Names: 2-CdA; 2CDA; CdA; Cladribina; Leustat; Leustatin; Leustatine; RWJ-26251
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Biological: Filgrastim — Given SC
  Other Names: FILGRASTIM, LICENSE HOLDER UNSPECIFIED; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim; Nivestym; Filgrastim-aafi
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Mitoxantrone — Given IV
  Other Names: Dihydroxyanthracenedione; Mitozantrone
Drug: Sorafenib — Given PO
  Other Names: 284461-73-0; BAY 43-9006; Bay-439006

SUMMARY:
This phase I/II trial studies the side effects and best dose of filgrastim (granulocyte colony-stimulating factor [G-CSF]), cladribine, cytarabine, and mitoxantrone, when given together with sorafenib and to see how well they work in treating patients with newly-diagnosed acute myeloid leukemia or high-risk myelodysplastic syndrome (likely to be more aggressive). Drugs used in chemotherapy, such as cladribine, cytarabine, and mitoxantrone work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Colony-stimulating factors, such as filgrastim, may increase the production of blood cells and may help the immune system recover from the side effects of chemotherapy. Sorafenib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving filgrastim, cladribine, cytarabine, and mitoxantrone together with sorafenib may kill more cancer cells.

DETAILED DESCRIPTION:
OUTLINE: This is a phase I, dose-escalation study of mitoxantrone and sorafenib followed by a phase II study.

INDUCTION: Patients receive mitoxantrone intravenously (IV) over 60 minutes on days 1-3 and sorafenib orally (PO) twice daily (BID) on days 10-19 in the absence of disease progression or unacceptable toxicity. Patients also receive filgrastim subcutaneously (SC) once daily (QD) on days 0-5, cladribine IV QD over 2 hours on days 1-5, and cytarabine IV QD over 2 hours on days 1-5 in the absence of disease progression or unacceptable toxicity. Patients achieving partial remission (including MRD positive [pos] CR, CR with incomplete platelet recovery [CRp], and CR with incomplete count recovery [CRi]) or persistent AML may receive up to 2 cycles of induction therapy per the discretion of the treating physician.

POST-REMISSION: Patients receive sorafenib PO BID on days 8-27 or 3 days prior to next cycle of treatment, whichever occurs first. Patients also receive filgrastim subcutaneously SC QD on days 0-5, cladribine IV QD over 2 hours on days 1-5, and cytarabine IV QD over 2 hours on days 1-5 in the absence of disease progression or unacceptable toxicity. Patients achieving MRDneg CR may receive up to 4 cycles of post-remission therapy. Patients achieving disease response (MRDpos CR, CRi/CRp, or persistent disease) may receive up to two induction cycles and 1 cycle of post-remission therapy with mitoxantrone omitted in cycle 3. If they then enter MRDneg CR, they can proceed with up to a total of 4 cycles of post-remission therapy.

MAINTENANCE THERAPY: Patients achieving MRDneg CR may receive maintenance therapy of sorafenib PO BID for up to 1 year.

After completion of study treatment, patients are followed up every 3 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years, inclusive
* Newly diagnosed disease with either a diagnosis of "high-risk" MDS (>= 10% blasts in marrow or blood), high-risk myeloproliferative neoplasm (MPN; >= 10% blasts in blood or bone marrow), or AML other than acute promyelocytic leukemia (APL) with t(15;17)(q22;q12) or variants according to the 2008 World Health Organization (WHO) classification. Patients with biphenotypic AML are eligible; such "high-risk" MDS or MPN have natural history much closer to AML than to lower risk MDS or MPN and have responded similarly to "AML-type" therapy.
* Outside diagnostic material is acceptable as long as peripheral blood and/or bone marrow slides are reviewed at the study institution by appropriate clinical staff. Flow cytometric analysis of peripheral blood and/or bone marrow should be performed according to institutional practice guidelines.
* Treatment-related mortality (TRM) score =< 13.1 as calculated with simplified model
* The use of hydroxyurea prior to study registration is allowed. Patients with symptoms/signs of hyperleukocytosis, white blood cell (WBC) > 100,000/uL, or acute symptoms can be treated with leukapheresis or may receive up to 2 doses of cytarabine (up to 500 mg/m^2/dose) prior to study day 0 enrollment
* Bilirubin =< 2 times institutional upper limit of normal unless elevation is thought to be due to hepatic infiltration by AML, Gilbert's syndrome, or hemolysis (assessed within 10 days prior to study day 0)
* Serum creatinine =< 2.0 mg/dL (assessed within 10 days prior to study day 0)
* Left ventricular ejection fraction >= 45%, assessed within 3 months prior to study day 0, e.g. by multi gated acquisition scan (MUGA) scan or echocardiography, or other appropriate diagnostic modality and no clinical evidence of congestive heart failure
* Women of childbearing potential and men must agree to use adequate contraception beginning at the signing of the consent until at least 3 months after the last dose of study drug
* Provide written informed consent (or legal representative)

Exclusion Criteria:

* Myeloid blast crisis of chronic myeloid leukemia (CML), unless patient is not considered candidate for CML-directed tyrosine kinase inhibitor treatment (excluding sorafenib)
* Concomitant illness associated with a likely survival of < 1 year
* Active systemic fungal, bacterial, viral, or other infection, unless disease is under treatment with anti-microbials and/or controlled or stable (e.g. if specific, effective therapy is not available/feasible or desired [e.g. chronic viral hepatitis, human immunodeficiency virus (HIV)]). Patient needs to be clinically stable as defined as being afebrile and hemodynamically stable for 24-48 hours prior to study day 0, unless fever is thought to be secondary to the underlying hematologic disease.
* Active or clinically significant (or symptomatic) cardiac disease, including active coronary artery disease, cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin within the last 3 months, unstable angina (anginal symptoms at rest), new-onset angina within 3 months before randomization, or myocardial infarction within 6 months before study day 0
* Previous receipt of azacitidine, decitabine, anthracyclines, cytarabine, or other nucleoside analogues for treatment of AML or MPN/MDS other than as noted for cytarabine
* Pregnancy or lactation
* Concurrent treatment with any other investigational agent that has anti-leukemia activity or another drug with anti-AML-activity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2023-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Halpern, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Halpern AB, Rodriguez-Arboli E, Othus M, Garcia KA, Percival MM, Cassaday RD, Oehler VG, Becker PS, Appelbaum JS, Abkowitz JL, Orozco JJ, Keel SB, Hendrie PC, Scott BL, Ghiuzeli MC, Estey EH, Walter RB. Phase 1/2 study of sorafenib added to cladribine, high-dose cytarabine, G-CSF, and mitoxantrone in untreated AML. Blood Adv. 2023 Sep 12;7(17):4950-4961. doi: 10.1182/bloodadvances.2023010392. PMID 37339483

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1, Dose Level 1: Sorafenib 200mg PO BID days 10-19 Mitoxantrone 10mg/m^2 IV days 1-3 G-CSF SQ 5µcg/kg days 0-5 Cladribine IV 5mg/m^2 days 1-5 Cytarabine IV 2g/m^2 days 1-5
- Phase 1, Dose Level 2: Sorafenib 200mg PO BID days 10-19 Mitoxantrone 12mg/m^2 IV days 1-3 G-CSF SQ 5µcg/kg days 0-5 Cladribine IV 5mg/m^2 days 1-5 Cytarabine IV 2g/m^2 days 1-5
- Phase 1, Dose Level 3: Sorafenib 200mg PO BID days 10-19 Mitoxantrone 15mg/m^2 IV days 1-3 G-CSF SQ 5µcg/kg days 0-5 Cladribine IV 5mg/m^2 days 1-5 Cytarabine IV 2g/m^2 days 1-5
- Phase 1, Dose Level 4: Sorafenib 200mg PO BID days 10-19 Mitoxantrone 18mg/m^2 IV days 1-3 G-CSF SQ 5µcg/kg days 0-5 Cladribine IV 5mg/m^2 days 1-5 Cytarabine IV 2g/m^2 days 1-5
- Phase 1, Dose Level 5: Sorafenib 400mg AM, 200mg PM PO days 10-19 Mitoxantrone 18mg/m^2 IV days 1-3 G-CSF SQ 5µcg/kg days 0-5 Cladribine IV 5mg/m^2 days 1-5 Cytarabine IV 2g/m^2 days 1-5
- Phase 1, Dose Level 6; Phase 2, Dose Level 6: Sorafenib 400mg PO BID days 10-19 Mitoxantrone 18mg/m^2 IV days 1-3 G-CSF SQ 5µcg/kg days 0-5 Cladribine IV 5mg/m^2 days 1-5 Cytarabine IV 2g/m^2 days 1-5
Period: Overall Study
Arm/Group | Phase 1, Dose Level 1 | Phase 1, Dose Level 2 | Phase 1, Dose Level 3 | Phase 1, Dose Level 4 | Phase 1, Dose Level 5 | Phase 1, Dose Level 6 | Phase 2, Dose Level 6
Started | 6 | 6 | 11 | 8 | 9 | 7 | 37
Completed | 6 | 6 | 11 | 8 | 9 | 7 | 37
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1, Dose Level 1 | Phase 1, Dose Level 2 | Phase 1, Dose Level 3 | Phase 1, Dose Level 4 | Phase 1, Dose Level 5 | Phase 1, Dose Level 6 | Phase 2, Dose Level 6 | Total
Number analyzed (Participants) | 6 | 6 | 11 | 8 | 9 | 7 | 37 | 84
Age, Customized [Median (Full Range); unit: years] | 40.5 [26 to 55] | 49.5 [24 to 53] | 41 [22 to 59] | 49 [35 to 59] | 56 [30 to 59] | 48 [23 to 57] | 49 [21 to 60] | 48 [21 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 6 | 7 | 4 | 5 | 11 | 38
  Male | 5 | 2 | 5 | 1 | 5 | 2 | 26 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 6 | 1 | 1 | 0 | 0 | 2 | 11
  Not Hispanic or Latino | 5 | 0 | 10 | 7 | 9 | 7 | 35 | 73
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 4
  Asian | 1 | 2 | 0 | 0 | 0 | 1 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3
  White | 4 | 2 | 8 | 8 | 8 | 5 | 30 | 65
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Disease classification [Count of Participants; unit: Participants]
  AML | 5 | 4 | 11 | 6 | 7 | 7 | 29 | 69
  MDS | 1 | 2 | 0 | 2 | 2 | 0 | 5 | 12
  CMML-2 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
MRC Risk Category [Count of Participants; unit: Participants]
  Favorable | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 5
  Intermediate | 4 | 5 | 8 | 6 | 7 | 6 | 24 | 60
  Adverse | 2 | 1 | 2 | 2 | 2 | 0 | 10 | 19
ELN 2017 Risk Group [Count of Participants; unit: Participants]
  Favorable | 2 | 2 | 4 | 0 | 5 | 2 | 10 | 25
  Intermediate | 0 | 2 | 2 | 5 | 0 | 4 | 13 | 26
  Adverse | 4 | 2 | 5 | 3 | 3 | 1 | 14 | 32
  Unable to assess | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Secondary Disease [Count of Participants; unit: Participants]
  Secondary disease | 0 | 0 | 1 | 5 | 0 | 0 | 7 | 13
  No secondary disease | 6 | 6 | 10 | 3 | 9 | 7 | 30 | 71
ECOG Performance Status [Count of Participants; unit: Participants] — 0: Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 2 | 1 | 0 | 2 | 2 | 1 | 2 | 10
    1 | 4 | 5 | 9 | 5 | 7 | 6 | 32 | 68
    2 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 5
    3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Treatment Related Mortality (TRM) Score [Median (Full Range); unit: units on a scale] — Our institution defines treatment-related mortality (TRM) as death within 28 days from initiation of chemotherapy based on observation that risk of death declines once 4 weeks has elapsed from treatment start. Calculation is used to predict TRM (scale from 0-100) using age, performance status, if they have secondary AML, albumin, creatinine, platelet count, white blood cell count, and peripheral blood blast percentage. The higher the TRM score, the higher the risk of TRM. Calculator and table of relationship between TRM score and TRM probability found here https://trmcalculator.fredhutch.org/
  units on a scale | 1.15 [0.20 to 2.83] | 2.00 [1.06 to 4.19] | 2.72 [0.6 to 7.2] | 2.19 [1.2 to 12.26] | 1.57 [0.56 to 2.28] | 1.28 [0.19 to 5.56] | 2.21 [0.26 to 8.42] | 1.96 [0.19 to 12.26]
FLT3 Mutations [Count of Participants; unit: Participants] — Mutations in FLT3 are the most common genetic alteration in AML. The FLT3 gene provides instructions for making a protein called fms-like tyrosine kinase 3 (FLT3). Two basic categories of mutation are recognized in FLT3: (1) FLT3-ITD, internal tandem duplication (ITD) within the FLT3 juxtamembrane domain and (2) FLT3-TKD, activating missense mutations affecting the tyrosine kinase domain (TKD).
  Participants
    FLT3-ITD mutation | 0 | 2 | 2 | 2 | 2 | 3 | 10 | 21
    FLT3-TKD mutation | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 6
    No FLT3 mutations | 4 | 3 | 8 | 5 | 6 | 2 | 24 | 52
    FLT3 mutation status unknown | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Maximum Tolerated Dose (MTD)/Recommended Phase 2 Dose (RP2D) of Mitoxantrone
Description: MTD/RP2D will be defined as the highest dose studied in which the incidence of dose-limiting toxicity (DLT) is < 33% assuming at least 6 patients have been treated at this dose. DLTs were defined as: 1) grade ≥3 non-hematologic toxicity lasting >48 hours leading to >7-day delay of the next cycle; 2) grade ≥4 non-hematologic toxicity if no recovery to grade ≤2 in 14 days (both excluding febrile neutropenia/ infection); 3) Absolute neutrophil count <500/ µL or platelet count <50,000/µL for >49 days after CLAGM+S without marrow evidence of AML. Doses were escalated up to dose level six if <2/6 patients out of each cohort of 6 had a DLT (some cohorts were expanded to 12 patients while awaiting completion of DLT monitoring period). The dose level at which dose escalation was stopped was the recommended phase 2 dose (RP2D).
Time Frame: First 28 days of treatment
Measure: Number; unit: mg/m^2
Groups:
- CLAGM+Sorafenib Phase 1: Participants enrolled during Phase 1 were assigned to one of six escalating dose levels. Six to 12 participants were enrolled in each dose level. Doses were escalated up to dose level 6 if <2 out of 6 participants out of each cohort had a dose limiting toxicity (DLT). The dose level at which dose escalation was stopped was the recommended phase 2 dose (RP2D).
Arm/Group | CLAGM+Sorafenib Phase 1
Number analyzed (Participants) | 47
mg/m^2 | 18

2. Primary Outcome: Phase 1: Maximum Tolerated Dose (MTD)/Recommended Phase 2 Dose (RP2D) of Sorafenib
Description: as for outcome 1
Time Frame: First 28 days of treatment
Measure: Number; unit: mg BID
Arm/Group | CLAGM+Sorafenib Phase 1
Number analyzed (Participants) | 47
mg BID | 400

3. Primary Outcome: Phase I and II: Rate of Minimal Residual Disease Negative (MRDneg) Complete Response (CR)
Description: We will determine if the addition of sorafenib to CLAG-M improves the rate of MRDneg CR compared to our institution's historical control of CLAG-M alone in adults with newly-diagnosed AML/high-risk MDS.
Time Frame: 56 days (2 cycles of induction chemotherapy)
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1, Dose Level 1: Sorafenib 200mg PO BID days 10-19 Mitoxantrone 10mg/m^2 IV days 1-3 G-CSF SQ 5µcg/kg days 0-5 Cladribine IV 5mg/m2 days 1-5 Cytarabine IV 2g/m2 days 1-5
- Phase 1, Dose Level 2: Sorafenib 200mg PO BID days 10-19 Mitoxantrone 12mg/m^2 IV days 1-3 G-CSF SQ 5µcg/kg days 0-5 Cladribine IV 5mg/m2 days 1-5 Cytarabine IV 2g/m2 days 1-5
- Phase 1, Dose Level 3: Sorafenib 200mg PO BID days 10-19 Mitoxantrone 15mg/m^2 IV days 1-3 G-CSF SQ 5µcg/kg days 0-5 Cladribine IV 5mg/m2 days 1-5 Cytarabine IV 2g/m2 days 1-5
- Phase 1, Dose Level 4: Sorafenib 200mg PO BID days 10-19 Mitoxantrone 18mg/m^2 IV days 1-3 G-CSF SQ 5µcg/kg days 0-5 Cladribine IV 5mg/m2 days 1-5 Cytarabine IV 2g/m2 days 1-5
- Phase 1, Dose Level 5: Sorafenib 400mg AM, 200mg PM PO days 10-19 Mitoxantrone 18mg/m^2 IV days 1-3 G-CSF SQ 5µcg/kg days 0-5 Cladribine IV 5mg/m2 days 1-5 Cytarabine IV 2g/m2 days 1-5
- Phase 1, Dose Level 6; Phase 2, Dose Level 6: Sorafenib 400mg PO BID days 10-19 Mitoxantrone 18mg/m^2 IV days 1-3 G-CSF SQ 5µcg/kg days 0-5 Cladribine IV 5mg/m2 days 1-5 Cytarabine IV 2g/m2 days 1-5
Arm/Group | Phase 1, Dose Level 1 | Phase 1, Dose Level 2 | Phase 1, Dose Level 3 | Phase 1, Dose Level 4 | Phase 1, Dose Level 5 | Phase 1, Dose Level 6 | Phase 2, Dose Level 6
Number analyzed (Participants) | 6 | 6 | 11 | 8 | 9 | 7 | 37
Participants | 3 | 6 | 8 | 4 | 9 | 7 | 31
Statistical Analysis 1: Comparison: Phase 1, Dose Level 1 vs Phase 1, Dose Level 2 vs Phase 1, Dose Level 3 vs Phase 1, Dose Level 4 vs Phase 1, Dose Level 5 vs Phase 1, Dose Level 6 vs Phase 2, Dose Level 6; Participants on study receiving CLAGM-S were compared to a historical cohort of newly diagnosed AML/high-risk MDS patients treated with CLAG-M alone, matched for mitoxantrone dose, age, and TRM score. Number of participants in historical cohort = 71. Number of participants in historical cohort who achieved MRD-negative CR = 55 (77.46%); Test type: Superiority; p = 0.48, Fisher Exact

4. Secondary Outcome: Complete Remission (CR)
Description: Complete remission (CR) is defined as bone marrow blasts <5%; absence of circulating blasts; absence of extramedullary disease; ANC ≥1.0 x 10^9/L; platelet count ≥100 x 10^9/L.
  CR with incomplete hematologic recovery (CRi) is CR with ANC <1.0 x10^9/L or platelet count <100 x 10^9/L.
  Measurable residual disease (MRD) is assessed by multiparameter flow cytometry and PCR.
  Morphologic leukemia free state (MLFS) is bone marrow blasts <5%; absence of circulating blasts; absence of extramedullary disease; no hematologic recovery.
  Resistant disease is defined as not not meeting the criteria for CR, CRi, MLFS.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1, Dose Level 1: Sorafenib 200mg PO BID days 10-19 Mitoxantrone 10mg/m2 IV days 1-3 G-CSF SQ 5µcg/kg days 0-5 Cladribine IV 5mg/m2 days 1-5 Cytarabine IV 2g/m2 days 1-5
- Phase 1, Dose Level 2: Sorafenib 200mg PO BID days 10-19 Mitoxantrone 12mg/m2 IV days 1-3 G-CSF SQ 5µcg/kg days 0-5 Cladribine IV 5mg/m2 days 1-5 Cytarabine IV 2g/m2 days 1-5
- Phase 1, Dose Level 3: Sorafenib 200mg PO BID days 10-19 Mitoxantrone 15mg/m2 IV days 1-3 G-CSF SQ 5µcg/kg days 0-5 Cladribine IV 5mg/m2 days 1-5 Cytarabine IV 2g/m2 days 1-5
- Phase 1, Dose Level 4: Sorafenib 200mg PO BID days 10-19 Mitoxantrone 18mg/m2 IV days 1-3 G-CSF SQ 5µcg/kg days 0-5 Cladribine IV 5mg/m2 days 1-5 Cytarabine IV 2g/m2 days 1-5
- Phase 1, Dose Level 5: Sorafenib 400mg AM, 200mg PM PO days 10-19 Mitoxantrone 18mg/m2 IV days 1-3 G-CSF SQ 5µcg/kg days 0-5 Cladribine IV 5mg/m2 days 1-5 Cytarabine IV 2g/m2 days 1-5
- Phase 1, Dose Level 6; Phase 2, Dose Level 6: Sorafenib 400mg PO BID days 10-19 Mitoxantrone 18mg/m2 IV days 1-3 G-CSF SQ 5µcg/kg days 0-5 Cladribine IV 5mg/m2 days 1-5 Cytarabine IV 2g/m2 days 1-5
Arm/Group | Phase 1, Dose Level 1 | Phase 1, Dose Level 2 | Phase 1, Dose Level 3 | Phase 1, Dose Level 4 | Phase 1, Dose Level 5 | Phase 1, Dose Level 6 | Phase 2, Dose Level 6
Number analyzed (Participants) | 6 | 6 | 11 | 8 | 9 | 7 | 37
Participants
  CR: MRD-negative | 3 | 6 | 8 | 4 | 9 | 7 | 31
  CR: MRD-positive | 2 | 0 | 0 | 0 | 0 | 0 | 1
  CRi: MRD-negative | 1 | 0 | 0 | 1 | 0 | 0 | 1
  CRi: MRD-positive | 0 | 0 | 0 | 0 | 0 | 0 | 1
  MLFS | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Resistant disease | 0 | 0 | 1 | 3 | 0 | 0 | 2
  Indeterminate | 0 | 0 | 0 | 0 | 0 | 0 | 1

5. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR, defined as CR+CRi, rates of patients treated with CLAG-M with sorafenib.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Dose Level 1 | Phase 1, Dose Level 2 | Phase 1, Dose Level 3 | Phase 1, Dose Level 4 | Phase 1, Dose Level 5 | Phase 1, Dose Level 6 | Phase 2, Dose Level 6
Number analyzed (Participants) | 6 | 6 | 11 | 8 | 9 | 7 | 37
Participants | 6 | 6 | 8 | 5 | 9 | 7 | 34

6. Secondary Outcome: Overall Survival (OS)
Description: 12-month overall survival
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Groups:
- CLAGM+Sorafenib Phase 2: Participants enrolled during phase 2 and treated at the recommended phase 2 dose that was established in phase 1. Patients treated at the RP2D in the Phase 1 were included in the Phase 2 analysis.
Arm/Group | CLAGM+Sorafenib Phase 2
Number analyzed (Participants) | 44
percentage of participants | 86

7. Secondary Outcome: Event-free Survival (EFS)
Description: 12-month event free survival
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | CLAGM+Sorafenib Phase 2
Number analyzed (Participants) | 44
percentage of participants | 81

8. Secondary Outcome: Relapse-free Survival (RFS)
Description: 12-month relapse free survival (RFS)
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | CLAGM+Sorafenib Phase 2
Number analyzed (Participants) | 44
percentage of participants | 82

9. Secondary Outcome: Number of Participants With Adverse Events
Description: Will be assessed using National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1, Dose Level 1 | Phase 1, Dose Level 2 | Phase 1, Dose Level 3 | Phase 1, Dose Level 4 | Phase 1, Dose Level 5 | Phase 1, Dose Level 6 | Phase 2, Dose Level 6
Number analyzed (Participants) | 6 | 6 | 11 | 8 | 9 | 7 | 37
Participants | 6 | 6 | 11 | 8 | 9 | 7 | 32

ADVERSE EVENTS:
Time Frame: From time of consent until 60 days after day 1 of each cycle, up to 5 years. Subjects can receive up to five cycles of therapy. After that, eligible subjects can receive maintenance therapy for up to one year. All-cause mortality was assessed for up to 5 years.
Arm/Group | Phase 1, Dose Level 1 | Phase 1, Dose Level 2 | Phase 1, Dose Level 3 | Phase 1, Dose Level 4 | Phase 1, Dose Level 5 | Phase 1, Dose Level 6 | Phase 2, Dose Level 6
All-Cause Mortality (participants affected / at risk) | 2/6 | 2/6 | 2/11 | 4/8 | 3/9 | 0/7 | 10/37
Serious Adverse Events (participants affected / at risk) | 2/6 | 2/6 | 4/11 | 4/8 | 4/9 | 5/7 | 22/37
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 10/11 | 8/8 | 8/9 | 6/7 | 27/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Dose Level 1 (N=6) | Phase 1, Dose Level 2 (N=6) | Phase 1, Dose Level 3 (N=11) | Phase 1, Dose Level 4 (N=8) | Phase 1, Dose Level 5 (N=9) | Phase 1, Dose Level 6 (N=7) | Phase 2, Dose Level 6 (N=37)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sweet's Syndrome (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (5) | 2 (6) | 3 (5) | 5 (5) | 16 (27)
GI malignancy (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perianal abscess (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Line associated DVT (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (10)
Sepsis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizire (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Dose Level 1 (N=6) | Phase 1, Dose Level 2 (N=6) | Phase 1, Dose Level 3 (N=11) | Phase 1, Dose Level 4 (N=8) | Phase 1, Dose Level 5 (N=9) | Phase 1, Dose Level 6 (N=7) | Phase 2, Dose Level 6 (N=37)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (9) | 6 (13) | 9 (14) | 7 (13) | 6 (8) | 2 (2) | 12 (45)
Bacteremia (Blood and lymphatic system disorders) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fever (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 6 (7) | 4 (4) | 7 (8)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac troponin I increased (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Edema face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toe infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Tongue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
C.difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injury to jugular vein (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was limited by its single-institution and non-randomized nature

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT02728050/Prot_SAP_000.pdf